CLINICAL TRIAL: NCT03689933
Title: Stability of Patient-specific Root-analogue Implants and Conventional Root-form Implants for Treating Non-restorable Single-rooted Maxillary Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr mohamed ahmed, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28902050100374
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Implant Stability; Root Analog Implant; Conventional Root Form Implant; Non Restorabl Teeth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- root analog implant (Experimental): The tooth indicated for extraction will be extracted atraumatically using periotome, socket preservation using Iodoform packing strips, and then optical scanning of the remaining tooth structure with optical scanner will be made to obtain a 3D virtual model, this model will be modified by addition of macro-retentions strictly to the interdental area to avoid any fracture in thin cortical bone, the cervical portion of implant circumference will be decreased by 0.1 to 0.2 mm to avoid pressure resorption of alveolar crest of bone and addition of prepared crown stump for the future crown to be placed.
  Interventions: Device: Root analog implant
- conventional stock root-form titanium implant (Active Comparator): Using a conventional implant as a comparator as it's the gold stander in restoring the non-restorable teeth.
  Interventions: Device: Root analog implant

INTERVENTIONS:
Device: Root analog implant — a custom made root analogue implant made from milled titanium
  Other Names: patient specific implant

SUMMARY:
its a experimental study comparing between the stability of immediate root fomed implant versus the conventional titanium implant

DETAILED DESCRIPTION:
Patients will be selected from the out-patient clinic according to the inclusion and exclusion criteria, from where the participants will be divided into two equal groups using computer generated random table and the sequence of the random numbers will be only revealed to the Co-supervisor who will report the assigned treatment to the principal investigator.

Immediate placement of root analogue titanium dental implants. All patients in the study group will be radiographed using cone beam computed tomography for diagnosis and evaluating the attachment of the tooth and bone level.

The tooth indicated for extraction will be extracted atraumatically using periotome, socket preservation using Iodoform packing strips, and then optical scanning of the remaining tooth structure with optical scanner will be made to obtain a 3D virtual model, this model will be modified by addition of macro-retentions strictly to the interdental area to avoid any fracture in thin cortical bone, the cervical portion of implant circumference will be decreased by 0.1 to 0.2 mm to avoid pressure resorption of alveolar crest of bone and addition of prepared crown stump for the future crown to be placed.

After all additions and adjustments are being made, an STL (stereolithography) extension file followed by milling of the implant from medically grade titanium will be carried out, followed by sandblasting acid etching.

For sterilization, the implant will be washed in a 90% concentration ethanol ultrasonic bath for 10 minutes, followed by packaging and sterilizing in a steam pressure autoclave.

At the day of implant placement, removing of suture and the Iodoform gauze followed by flushing of the extraction socket using saline solution and vigorous curettage of the socket. Then implant placement will be made by hand pressure followed by tapping using mallet.

Implant stability in both groups will be measured using Periotest device. The measuring procedure will be made immediate postoperative, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Single rooted teeth indicated for extraction and immediate implant placement.
2. The age of candidates ranges from 21 to 50 years.

Exclusion Criteria:

1. Absence of any disease or systemic complication which might affect osseointegration.
2. The cause of extraction mustn't be due to periodontitis or periapical infection.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
implant stability | 6 months
  using periotest

IPD SHARING:
Plan to Share IPD: Undecided